CLINICAL TRIAL: NCT04964479
Title: A Randomized, Blind, Parallel Controlled, Multicenter Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsules Versus Pembrolizumab Injection as a First-line Treatment on Patient With Advanced NSCLC.
Brief Title: A Clinical Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsules Versus K Drug in the Treatment of First-line Non-small Cell Lung Cancer(NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TQB2450-III-09
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 injection + Anlotinib Hydrochloride capsules (Experimental): TQB2450 injection: once every 3 weeks, 1200mg each time, intravenous infusion. Until the disease progression or unbearable adverse events occur.
  Anlotinib Hydrochloride capsules: once a day,12mg each time, oral administration before breakfast. Continuous administration for 2 weeks, withdrawal for 1 week, i.e. 3 weeks (21 days) as a course of treatment. Until the disease progression or unbearable adverse events occur.
  Interventions: Drug: TQB2450 injection; Drug: Anlotinib Hydrochloride Capsules
- Pembrolizuma injection + placebo of Anlotinib hydrochloride capsules (Active Comparator): Pembrolizumab injection: once every 3 weeks, 200mg each time, intravenous infusion. Until the disease progression or unbearable adverse events occur.
  Placebo of Anlotinib hydrochloride capsules:once a day, 0mg each time, oral administration before breakfast. Continuous administration for 2 weeks, withdrawal for 1 week, i.e. 3 weeks (21 days) as a course of treatment. Until the disease progression or unbearable adverse events occur.
  Interventions: Drug: Pembrolizumab injection; Drug: Placebo

INTERVENTIONS:
Drug: TQB2450 injection — 1200mg injection once every 3 week
  Arms: TQB2450 injection + Anlotinib Hydrochloride capsules
Drug: Anlotinib Hydrochloride Capsules — 12mg capsule once daily
  Arms: TQB2450 injection + Anlotinib Hydrochloride capsules
Drug: Pembrolizumab injection — 200mg injection once every 3 week
  Arms: Pembrolizuma injection + placebo of Anlotinib hydrochloride capsules
Drug: Placebo — Placebo capsule once daily
  Arms: Pembrolizuma injection + placebo of Anlotinib hydrochloride capsules

SUMMARY:
A clinical study to evaluate the efficacy and safety of TQB2450 injection combined with Anlotinib Hydrochloride capsules versus K drug as a first-line treatment of advanced non-small cell lung cancer.A total of 375 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* According to the 8th edition of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification, the tumor node metastasis (TNM) staging of lung cancer is locally advanced (stage ⅢB/ⅢC), metastatic or recurrent ( Stage IV) NSCLC patients. (Note: Mixed tumors will be classified according to the main cell type; if there are small cell components, the subject is unqualified).
* Between the ages of 18-75 years (calculated based on the date of signing ICF); male or female; Eastern cooperative oncology group (ECOG) score 0-1; estimated survival time ≥ 3 months.
* According to the RECIST 1.1 standard, there is at least one measurable lesion. If the measurable lesion is located in the radiotherapy area, it should be clearly defined as a progressive state.
* Patients who have not received systemic anti-tumor therapy for advanced, recurrent or metastatic diseases in the past. For those who have received adjuvant chemotherapy in the past, the interval between the recurrence time and the last adjuvant chemotherapy should be at least 6 months; The interval between the end of previous radiotherapy for chest and this treatment should be more than 6 months, and the interval between palliative radiotherapy for chest and this treatment should be more than 7 days.
* Tumor tissue slices that have not undergone radiotherapy at or after the diagnosis of advanced or metastatic NSCLC must be provided. Tumor tissue samples must be archived samples or fresh samples obtained within 12 months before randomization, and the proportion of programmed death-Ligand 1(PD-L1) positive tumor cells≥ 1% (TPS ≥ 1%).
* For non-squamous NSCLC, patients with no epidermal growth factor receptor (EGFR) mutations and ALK fusions (for squamous NSCLC, patients with known EGFR mutations and anaplastic Lymphoma kinase (ALK) fusions need to be excluded, and those with unknown status are not mandatory to be tested).
* The function of main organs are well and meet the following standards:

  a. Routine blood examination standards (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days before screening): i. Absolute neutrophil count (ANC) ≥1.5×109 /L; ii. Platelets ≥100×109 /L; iii. Hemoglobin ≥90 g/L. b. The blood biochemical examination shall meet the following standards: i. Total bilirubin (TBIL) ≤ 2 × upper limit of normal (ULN) (Patients with Gilbert syndrome ≤ 3 × ULN); ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN. If it is accompanied by liver metastasis, ALT and AST≤5×ULN; iii. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance estimated by Cockcroft-Gault glomerular filtration formula ≥60 mL/min; iv. Serum albumin (ALB) ≥30g/L. c. Urine routine examination standard: urine routine indicates urine protein <++; if urine protein ≥++, it is necessary to confirm that the 24-hour urine protein quantitative ≤1.0 g.

  d. Blood coagulation test standards: prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR)≤1.5×ULN (no anticoagulant therapy).

  e. Thyroid Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be examined. If T3 and T4 levels are normal, it can be selected.

  f. Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.

  g. 12-lead ECG evaluation: QTc<450ms (male), QTc<470ms (female).
* Women of childbearing age should agree to use effective contraceptive measures during the study period and 6 months after the end of the study, and have a negative serum pregnancy test within 7 days before the study enrollment; men should agree to the study period and 6 months after the end of the study period Effective contraceptive measures must be used internally.
* The subjects voluntarily joined the study, signed the informed consent form, and had good compliance.

Exclusion Criteria:

* Tumor disease and medical history:

  1. Brain metastases without local treatment; Note: Subjects who have previously received brain metastasis therapy and meet all the following criteria can participate in this study: i. Only supratentorial and cerebellar metastases; ii. The condition needs to be stable for ≥4 weeks and no new brain metastases or brain metastases are found Expanded imaging evidence; iii. The subject must have stopped corticosteroids/dehydrator for at least 2 weeks before starting to use the trial drug;
  2. There are midbrain, pons, medulla oblongata, spinal cord and meningeal metastases；
  3. Other malignant tumors appeared or were present within 3 years. The following two cases can be included: other malignant tumors treated by single operation have achieved 5-year Disease-free survival (DFS) in a row; The cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non-invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  4. Central type, cavity squamous cell carcinoma (primarily in the main bronchus and around the hilar);
  5. Imaging shows that the tumor invades large blood vessels or is unclearly separated from the blood vessels, or the investigator judges that the tumor is likely to invade important blood vessels and cause fatal bleeding during the subsequent study(The major vessels in the chest include pulmonary aorta, left pulmonary artery, right pulmonary artery, four pulmonary veins, superior vena cava, inferior vena cava and aorta);
  6. Severe bone injury caused by tumor bone metastasis, including pathological fracture of weight-bearing bone and spinal cord compression that occurred within 6 months or is expected to occur in the near future(Such as spine, pelvis, femur, tibia, phalanges, calcaneus, etc.);
  7. Patients with serous cavity (thoracic cavity, abdominal cavity, or pericardial cavity) that require repeated drainage to relieve clinical symptoms (as determined by the investigator), or who have received drainage of serous cavity effusion for the purpose of treatment within 2 weeks before treatment.
* Previous anti-tumor treatments:

  1. Received the treatment of proprietary Chinese medicines with anti-tumor indications specified in the NMPA approved drug instructions within 2 weeks before the start of the study treatment(Including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.);
  2. Previously received related immunotherapy drugs for programmed death 1 (PD-1), PD-L1, cytolytic T lymphocyte-associated antigen-4 (CTLA-4), etc.;
  3. Previous use of anti-angiogenic drugs such as bevacizumab, anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib, etc.;
  4. Patients who have been vaccinated with immunomodulatory drugs within 30 days before starting treatment(Such as interleukin-2, thymosin, lentinan, etc.);
  5. Failure to recover from the toxicity and/or complications of previous interventions to CTCAE ≤1, except for hair loss and peripheral neuropathy ≤2;
* Combined diseases and medical history:

  a. Liver cirrhosis, active hepatitis*;(Note: active hepatitis (hepatitis B reference: HBV-DNA > 1*103 copy /mL or > 2000IU/mL) when HBsAg is positive. Hepatitis C reference: HCV antibody is positive, and HCV titer detection value exceeds the upper limit of normal value); b. Renal abnormalities: i.Renal failure requires hemodialysis or peritoneal dialysis; ii.Previous or existing nephrotic syndrome, chronic nephritis. c. Cardiovascular and cerebrovascular abnormalities： i.Patients with previous or present heart failure, degree II or above heart block: ii.Myocardial infarction or unstable angina, supraventricular or ventricular arrhythmia with clinical significance need treatment or intervention; iii.Vascular embolism and cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage and cerebral infarction) occurred within 9 months（ Prophylactic use of anticoagulant therapy is allowed for patients with thrombotic tendency or undergoing anticoagulant therapy.) iv.After more than two kinds of drug treatment, blood pressure control is still not ideal (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg).

  d. Gastrointestinal abnormalities: i.Inability to take medications (such as inability to swallow, intestinal obstruction, etc.); ii.A history of malabsorption syndrome or other diseases that interfere with gastrointestinal absorption; iii.Received treatment for active peptic ulcer in the past 6 months; iv.Despite the maximum medical treatment, chronic diarrhea of grade 2 and above continues to occur; v.Other conditions determined by the researcher that may cause gastrointestinal bleeding and perforation.

  e. History of immunodeficiency: i.Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases; ii.Active autoimmune disease or history of autoimmune disease, including but not limited to Crohn's disease, ulcerative colitis, autoimmune hepatitis/enteritis/vasculitis/nephritis, etc.

iii.Prepare to undergo or have previously received an organ transplant; iv.Patients who require systemic or topical immunosuppressive therapy to achieve immunosuppressive purposes and need to continue to use them within two weeks before randomization (except for glucocorticoid daily dose <10 mg prednisone or other equivalent hormones).

Note: Hormone replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered as systemic therapy and allowed to be used.

f. Bleeding risk: i.Suffered from bleeding or coagulopathy within 28 days before the start of treatment or was using warfarin, aspirin and other antiplatelet agglutination drugs (except for aspirin ≤100 mg/d preventive drugs); ii.Had hemoptysis >2.5 mL/day in 28 days before the start of treatment; iii.Regardless of the severity, patients with any history of bleeding or coagulopathy; iv.Received major surgical treatment, open biopsy, etc. within 28 days before the start of the study treatment; v.Long-term unhealed wounds or fractures, except for pathological fractures; g. Poor control of type I diabetes or II diabetes (fasting blood glucose (FBG)> 10mmol/L); h. Severe infections within 4 weeks before the start of study treatment, including but not limited to hospitalization due to bacteremia, severe pneumonia, or other severe infections; subjects with ≥ grade 2 active infections within 4 weeks before the start of study treatment Or fever of unknown cause occurred during the screening period and before the first administration>38.0℃; i. Past or existing pneumoconiosis, interstitial pneumonia, (non-infectious) pneumonia that requires adrenal corticosteroid therapy, currently suffering from other types of pneumonia ≥2, or lung function tests confirmed severely impaired lung function (Forced Expiratory Volume in the first second (FEV1) or diffusing capacity of lung for carbon monoxide(DLCO) or DLCO per alveolar volume (DLCO /VA) accounts for the expected value %<40%) and other objective evidence; j. Patients with active tuberculosis within 1 year before enrollment; subjects with a history of active pulmonary tuberculosis infection 1 year ago must provide clear evidence of cure before enrollment; if tuberculosis is suspected during the screening period, chest radiographs and sputum must be passed Enter the group only after the liquid and clinical symptoms are eliminated; k. Allergies, or a history of severe allergies in the past, or severe hypersensitivity reactions after receiving other monoclonal antibody treatments, or known allergies to the ingredients of the study drug excipients; l. Previous history of severe mental disorders; m. People with a history of drug abuse, alcohol or drug abuse;

* The end of the previous clinical study (last dose) is less than 4 weeks or the study drug's 5 half-lives, whichever is shorter.
* Live attenuated vaccine vaccination history within 28 days before randomization or planned live attenuated vaccination during the study period. Seasonal influenza vaccine for injection is usually an inactivated virus vaccine and is allowed to be vaccinated during the study period.
* Female patients during pregnancy or lactation.
* According to the investigator's point of view, it may increase the risks associated with participating in the study, or other severe, acute or chronic medical diseases or laboratory abnormalities that may interfere with the interpretation of the study results, or other reasons that are not suitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival(PFS) evaluated by Independent Review Committee (IRC) | Baseline to up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first)

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline to up to two years
  The preriod from the first use of the drug to death from all causes. For subjects who are still alive at the last follow-up, the OS will be counted as data censored based on the last follow-up. For subjects who are lost follow-up, the OS will be counted as data censored based on the last confirmed survival time before being lost to follow-up.
Disease PFS evaluated by investigators | Baseline to up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first)
Objective response rate (ORR) evaluated by investigators | Baseline to up to two years
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and iRECIST, the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.
Disease Control Rate (DCR) | Baseline to up to two years
  Proportion of subjects whose tumors shrink or remain stable for a certain period, including CR, PR and stable disease（SD）
Duration of response (DOR) | Baseline to up to two years
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first) .
DOR rate (≥ 6 months) (the proportion of subjects with DOR ≥ 6 months) | Baseline to up to two years
  The proportion of subjects reaching 6 months from firstly- recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurred first) .
OS rate of 12 months | Baseline to up to two years
  The proportion of subjects who survive for 12 months after the first dose
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)，as well as abnormal laboratory examination indicators. | Baseline to up to two years
  The proportion of AEs and SAEs recorded afte signing the informed consent form(ICF).

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhangjiang, Guangdong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The Ninth Affiliated People's Hospital of Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Chongqing University, Chongqing
  - Three Gorges Hospital of Chongqing University, Chongqing
  - Southern Hospital of Southern Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The Fifth Central Hospital of Tianjin, Tianjin

REFERENCES:
- [Derived] Zhang W, Wang J, Wang Q, Cheng Y, Yang L, Li Y, Zhong H, Chu T, Dong Y, Zhang Y, Qian F, Xiong L, Shi C, Zhang C, He Z, Zhu J, Liu X, Ma H, Li K, Han B. A randomized double-blind trial of TQB2450 with or without anlotinib in pretreated driver-negative non-small cell lung cancer. Lung Cancer. 2023 Oct;184:107353. doi: 10.1016/j.lungcan.2023.107353. Epub 2023 Aug 21. PMID 37647728